CLINICAL TRIAL: NCT06192537
Title: Examining the Effect of Role-playing Exercise by Utilizing an Obesity Suit in a Simulation Scenario on Weight Bias and Empathy Levels Among Nutrition Sciences Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ariel University (Other)
Collaborators: Tel Hai College (Other)
Responsible Party: Principal Investigator, Shiri Sherf Dagan, Principal investigator, Ariel University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AU-HEA-SS-20231016-2
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Obesity; Bias, Weight
MeSH Terms: conditions — Obesity; Weight Prejudice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Behavioral: A role-playing exercise by utilizing an obesity suit in a simulation scenario

INTERVENTIONS:
Behavioral: A role-playing exercise by utilizing an obesity suit in a simulation scenario — All participants will be asked to wear an obesity simulation suit (Unisex obesity Simulation suit, Erler-Zimmer, Germany) and to participate in a standardized scenario that simulates meetings between a person with obesity and a 'registered dietitian'. The 'registered dietitian' will be presented by a professional role-player and the scenario will encompass different levels of weight bias through dialogue and the use of inappropriate equipment.

SUMMARY:
A quasi-experimental design (i.e., "One-Group Pretest-Posttest Design") will be applied among 34 convenient samples of undergraduate students in their first year of nutrition sciences program at Ariel University and Tel-Hai College. The intervention will take place at the simulation centers of the institutions. All participants will be asked to wear an obesity simulation suit (Unisex obesity Simulation suit, Erler-Zimmer, Germany) and to participate in a standardized scenario that simulates meetings between a person with obesity and a 'registered dietitian'. The 'registered dietitian' will be presented by a professional role-player and the scenario will encompass different levels of weight bias. At baseline, 1- and 3-week post-intervention both groups will be asked to fill in a survey using "Qualtrics" software. The survey will include the Anti-Fat Attitudes questionnaire (AFA), the Short-Form of Fat-Phobia scale (F-scale), the Weight-Implicit Association-Test (weight-IAT), and the Jefferson Scale of Empathy. Data on demographics, weight history, and perception, measurement of actual weight and height, and the beliefs about the causes of obesity questionnaire will be collected at baseline.

ELIGIBILITY:
Inclusion Criteria:

* undergraduate students in their first year of the nutrition sciences program at Ariel University or Tel-Hai College
* age ≥18 years
* having fluency in Hebrew
* ability to wear an obesity suit
* willingness to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Anti-Fat Attitudes questionnaire ('AFA') | Change from baseline at three- weeks post-intervention
  The 'AFA' indicates explicit anti-fat attitudes toward people with obesity and is composed of 13-items rated on a 10-point Likert scale and divided into three subscales ('dislike', 'fear about fat' and 'willpower'), with higher total scores indicating stronger anti-fat attitudes.
The short-form of fat-phobia scale (' F-scale') | Change from baseline at three- weeks post-intervention
  The 'F-scale' indicates fat-phobic attitudes toward people with obesity and is composed of 14-pairs of adjectives that are used to describe people with obesity (e.g., 'no willpower' vs. 'has willpower') and ranked on a 1-5 scale according to the point closest to the adjective name that describes their feelings and beliefs. Higher scores indicate stronger fat-phobic attitudes.
Weight Implicit Association Test ('IAT') | Change from baseline at three- weeks post-intervention
  IAT tool is an indirect measure of implicit bias toward weight which uses the constructs of "fat people" versus "thin people" and the polarized attitudes of "good" and "bad" to detect implicit weight bias.
The Jefferson Scale of Empathy (S-version) | Change from baseline at three- weeks post-intervention
  A 20-item scale that is designed to measure empathy in medical students.

SECONDARY OUTCOMES:
Demographics | At baseline
  Questions regarding age, gender, occupation, marital status, and religious affiliation.
Weight perception | At baseline
  Questions regarding self-definition of weight status, the importance of weight to self-confidence, and much control a person has over the weight.
Weight history | At baseline
  Questions regarding obesity during childhood, obesity during last decade, family members who struggle with obesity, currently in any process of losing weight.
Objective weight measurement | At baseline
  Measurement of actual weight in kilograms.
Objective height measurement | At baseline
  Measurement of actual height in meters.
The beliefs about the causes of obesity questionnaire | At baseline
  Rating the importance of 20 factors contributing to obesity by using a 5-point Likert-scale response format.

CONTACTS AND LOCATIONS:
Locations (1):
- Ariel University, Ariel, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tayar-Wachsberger I, Green G, Pinus M, Tepper S, Sherf-Dagan S. Examining the effect of an obesity suit role-playing exercise on empathy and weight bias in nutrition students. Nutrition. 2025 Oct;138:112813. doi: 10.1016/j.nut.2025.112813. Epub 2025 Apr 19. PMID 40466592